CLINICAL TRIAL: NCT04730843
Title: An Open-label, Multicenter, Dose-escalation and Cohort Expansion Phase 1 Clinical Study of ES102 Administered as a Single Agent in Patients With Advanced Solid Tumors
Brief Title: A Study of ES102 (OX40 Agonist) in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Elpiscience Biopharma, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ES102-1001
Record Dates: First submitted 2021-01-26; First posted 2021-01-29 (Actual); Last update posted 2025-06-23 (Actual); Status verified 2025-06

CONDITIONS: Solid Tumors; Neoplasms; Malignant Tumor
Keywords: ES102; solid tumor; phase 1; OX40; INBRX-106
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Part A dose escalation (Experimental): ES102 will be escalated in patients with advanced solid tumors.
  Interventions: Drug: ES102
- Part B expansion (Experimental): Subjects with advanced non-small cell lung cancer, advanced esophageal squamous cell carcinoma, other advanced solid tumors (such as nasopharyngeal carcinoma, cervical cancer, gastrointestinal tumors, other reproductive system tumors, etc.) will be treated with ES102 at the RP2D.
  Interventions: Drug: ES102

INTERVENTIONS:
Drug: ES102 — ES102 is administered via intravenous injection once every 21 days, every 21 days as a treatment cycle.

SUMMARY:
The purpose of this study is to evaluate the safety, tolerance, Dose-Limiting Toxicity (DLT), Maximum tolerated dose (MTD) and/or Recommended Phase 2 Dose (RP2D) of ES102 (OX40 Agonist) administered as a single agent in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and the willingness to sign a written informed consent form.
2. Males or females aged ≥18 years.
3. Part A: Subjects with pathological or cytological diagnosed advanced solid tumor, whose disease has progressed despite standard therapies, or for whom no further standard therapy exists, or who is unsuitable for available standard therapies.

   Part B: Subjects with NSCLC, ESCC, NPC, GI or Cervical cancers, with advanced disease, which has progressed despite all standard therapies or for whom no standard therapy exists, or who is unsuitable for available standard therapies.

   All subjects with NSCLC have documentation of absence of tumor activating EGFR mutation and absence of ALK and ROS1 gene rearrangements.
4. PD-L1 by IHC result mandatory but any score allowed .
5. At least one measurable lesion is required (RECIST v1.1)
6. Adequate hematologic, coagulation, hepatic and renal function as defined per protocol.
7. Eastern Cooperative Oncology Group performance status (ECOG PS) of 0 or 1.
8. Estimated life expectancy, in the judgment of the investigator, of at least 12 weeks.
9. Male and female subjects of childbearing potential and their spouses must be willing to use feasible contraceptive methods considered effective by the investigator, from the time of signing informed consent and for the duration of study participation through 3 months, following the last dose of study drug. Postmenopausal women are considered to have no fertility potential only if menostasis lasts for at least 12 months.

Exclusion Criteria:

1. Prior exposure to OX40 agonists.
2. Known allergies to CHO-produced antibodies, which in the opinion of the Investigator suggests an increased potential for an adverse hypersensitivity to ES102.
3. Receipt of any anticancer investigational product or any approved anticancer drug(s) or biological product(s) within 4 weeks prior to the first dose of study drug with certain exceptions.
4. Patients with other malignancies within 2 years before screening shall be excluded in Part B. Some exceptions as defined per protocol apply.
5. Hematologic malignancies (e.g., ALL, AML, MDS, CLL, CML, NHL, Hodgkin's lymphoma and multiple myeloma)
6. Known or active primary central nervous system (CNS) tumors, leptomeningeal disease and CNS metastases. Exception: subjects with previously treated, asymptomatic, and clinically stable CNS metastases may be allowed study entry if certain criteria apply in Part B.
7. Grade ≥ 3 immune-related adverse events (irAEs) or irAE that lead to discontinuation of prior immunotherapy. Some exceptions as defined per protocol apply.
8. Active autoimmune disease or documented history of autoimmune disease that required systemic steroids or other immunosuppressive medications. Certain exceptions as defined in protocol apply.
9. Treatment with systemic immunosuppressive medications within 4 weeks prior to the first dose of study drug. Certain exceptions as defined in protocol apply.
10. History of hepatitis B, hepatitis C, or human immunodeficiency virus (HIV) infection for Part A. Exceptions as defined in protocol for Part B will apply.
11. Active interstitial lung disease (ILD) or pneumonitis or a history of ILD or pneumonitis requiring treatment with steroids or other immunosuppressive medications.
12. Clinically significant cardiac condition, including myocardial infarction, uncontrolled angina, cerebrovascular accident, or other acute uncontrolled heart disease < 6 months; left ventricular ejection fraction (LVEF) < 50%; New York Heart Association (NYHA) Class III or IV congestive heart failure; or uncontrolled hypertension.
13. Active, hemodynamically significant pulmonary embolism within 3 months prior to the first dose of study drug.
14. Major surgery within 4 weeks prior to enrollment on this trial.
15. Systemic anti-infectious drug treatments within 4 weeks prior to the first dose of study drug.
16. Prior organ allograft transplantations or allogeneic peripheral blood stem cell (PBSC) or bone marrow (BM) transplantation.
17. Pregnant or nursing females.
18. Any known, documented, or suspected history of substance abuse that would preclude subject from participation, unless clinically justified (i.e., will not interfere with study participation and/or will not compromise trial objectives) per judgment of the Investigator and with approval of the Medical Monitor or Study Director.
19. The subject is inappropriate to participate in this study for other reasons in the judgment of the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) and/or Recommended Phase 2 Dose (RP2D) of of ES102 | 2-3 years
  The MTD and/or RP2D of ES102 will be determined.
Number of participants with adverse events and serious adverse events of ES102 | 2-3 years
  The safety profile of ES102 will be assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 5.0.

SECONDARY OUTCOMES:
Area under the serum concentration time curve (AUC) of ES102 | 2-3 years
  Area under the serum concentration time curve (AUC) of ES102 will be determined.
Maximum observed serum concentration (Cmax) of ES102 | 2-3 years
  Maximum observed serum concentration (Cmax) of ES102 will be determined.
Trough observed serum concentration (Ctrough) of ES102 | 2-3years
  Trough observed serum concentration (Ctrough) of ES102 will be determined.
Time to Cmax (Tmax) of ES102 | 2-3years
  Time to Cmax (Tmax) of ES102 will be determined.
Immunogenicity of ES102 | 2-3years
  Frequency of anti-drug antibodies (ADA) against ES102 will be determined.
Anti-tumor activity of ES102 | 2-3years
  Tumor response will be determined by the revised Response Evaluation Criteria in Solid Tumors version 1.1 (RECISTv1.1).

CONTACTS AND LOCATIONS:
Locations (1):
- Jilin Cancer Hospital, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No